CLINICAL TRIAL: NCT00881010
Title: Automated Pain Intervention for Underserved Minority Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0380; NCI-2012-02119 (Registry Identifier: NCI CTRP); RSGT-05-219-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Pain Intervention; Underserved minority patients; African American; Hispanic; Automated Telephone System for measuring symptoms; Interactive voice response; IVR
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telephone Intervention
  Interventions: Behavioral: Telephone Intervention; Behavioral: Questionnaires
- Usual Care
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Telephone Intervention — Automated Telephone Interactive Voice Response (IVR) system taking approximately 5 minutes, 2 times week for 10 weeks, to rate pain and symptoms.
  Groups: Telephone Intervention
Behavioral: Questionnaires — Surveys approximately 1 hour each at 2 regularly scheduled clinic visits to rate pain and symptoms. Regardless of group, all symptoms are to be reported.

SUMMARY:
The goal of this psychosocial research study is to learn about treating pain and other symptoms of minority patients who have breast cancer. The study will test how well a special telephone system works for improving the pain and symptom management of these patients.

DETAILED DESCRIPTION:
The special telephone system used in this study calls patients on a regular basis and asks them to report their symptoms. The patient's doctor or nurse is notified by a page or e-mail when one or more of these symptoms is severe: pain, shortness of breath, nausea, vomiting, drowsiness, sadness, and emotional distress. Researchers want to find out if using the telephone system is a better way to manage a patient's pain and symptoms than the normal method, in which the doctor and nurse would simply ask about pain and other symptoms.

You will be asked to complete several questionnaires during a visit to the oncology clinic. These questionnaires measure pain and other symptoms, quality of life, and mood. Completing the questionnaires takes about 1 hour. These will be completed during your first study visit (called the "baseline" visit.)

If you choose to take part in this study, you will be randomly assigned (as in the toss of a coin) to receive 1 of 2 treatment plans: telephone intervention or usual care. You have an equal chance of being assigned to either group.

If you are picked to be in the "telephone intervention" group, the research nurse will teach you how to use the telephone system for measuring symptoms. The research nurse also will ask you to practice using the telephone system. The telephone system will call you 2 times a week for 10 weeks and ask you to rate your pain and other symptoms and how much the symptoms interfere with your life. You can set up the most convenient times for the telephone calls. Rating your symptoms using the telephone system takes less than 5 minutes for each call.

Your symptom information from the telephone system will be given to your doctor and nurse at M. D. Anderson. The doctor or nurse will be notified right away by page or e-mail when one or more of these symptoms is severe: pain, shortness of breath, nausea, vomiting, drowsiness, sadness, and emotional distress. Patients in this group will also receive education from the telephone system about pain and pain treatments. If for some reason the telephone system is not working, the research staff will report your severe symptoms to your doctor of nurse, and give you the education about pain and pain treatments.

If you are assigned to the "usual care" group, then you will not be asked to report symptoms using the telephone system, and your symptom information from the questionnaires will not be given to your doctor and nurse at M. D. Anderson.

No matter what group you are assigned to, you will be asked to report all symptoms to your doctor and nurse during your visits to the oncology clinic. You will also be asked to call your doctor or nurse when symptoms are severe. The doctors and nurses will give you instructions about calling when your symptoms are severe.

You will be asked to fill out questionnaires during 2 regularly-scheduled clinic visits--at the visit 4-6 weeks after the study begins and at the visit 8-10 weeks after the study begins. These questionnaires measure pain and other symptoms, quality of life, and mood. Completing the questionnaires takes about 1 hour.

If you agree to participate in the companion caregiver study, the study staff will use your demographic and clinical data to study the influence of your symptoms on your caregiver's physical and mental health.

Your total participation in this study will be up to 10 weeks.

This is an investigational study. Up to 60 patients will take part in this multicenter study. About 10 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast cancer
2. African American or Hispanic female
3. Receiving treatment at LBJ General Hospital, Ben Taub Hospital, or M.D. Anderson Cancer Center
4. Socioeconomically disadvantaged, as indicated by hospital billing code
5. 18 years of age or older
6. Living in the United States
7. Speaks English or Spanish
8. "Pain worst" score of 4 or greater on the Brief Pain Inventory

Exclusion Criteria:

1. Current diagnosis of psychosis or dementia
2. No access to telephones
3. Unable to use the IVR system due to physical limitations (e.g., hearing impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disadvantaged African American or Hispanic females diagnosed with breast cancer aged 18 years or older with access to telephones.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-02 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
MDASI IVR Patient Symptom Assessment | Twice weekly

CONTACTS AND LOCATIONS:
Overall Officials: Tito Mendoza, PHD, MS, MED, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org